CLINICAL TRIAL: NCT05314465
Title: Effectiveness of Neural Mobilization on Spasticity and Upper Limb Function in Individuals With Stroke
Brief Title: Neural Mobilization for Reduction of Spasticity in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asir John Samuel (Other)
Responsible Party: Sponsor-Investigator, Asir John Samuel, Professor, Maharishi Markendeswar University (Deemed to be University)
Organization: Maharishi Markendeswar University (Deemed to be University) (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMDU/IEC/1935; U1111-1276-6515 (Other: WHO (UTN))
Record Dates: First submitted 2022-03-30; First posted 2022-04-06 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Stroke
Keywords: Stroke, spasticity, neural mobilization, Upper limb
MeSH Terms: conditions — Stroke; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Median nerve mobilization (Experimental): Experimental arm given Median nerve mobilization for 12mins 3sets for 3mins each with 1 minute interval in between for 5times a week for 4weeks
  Interventions: Other: Median nerve mobilization

INTERVENTIONS:
Other: Median nerve mobilization — Median nerve mobilization was given 20 oscillations per minute for 3 times & repeated 3 times with a pause of 1 minute between each sets for 5times/week for 4weeks.

SUMMARY:
Spasticity after stroke is common that affect upper limb strength and make activities of daily living difficult. There are many techniques but not any standardized technique for long term effect on reduction of spasticity and improving upper limb strength. This study aimed to explore and understand the effectiveness of neural mobilization on reduction of spasticity and improving upper limb strength in individuals with stroke. This is mixed method approach of embedded design, multicentric study recruited 7 individuals with stroke as no new themes or codes were emerging (data saturated). Median nerve mobilization was given 20 oscillations per minute for 3 times & repeated 3 times with a pause of 1 minute between each sets for 5times/week for 4weeks. Outcome measures were Modified Ashworth Scale (MAS), Brunnstrom's grading of hand recovery and Hydraulic hand dynamometer(HHD) for grip and pinch strength. Pre and post outcomes data were collected at baseline and 4weeks after intervention and in depth face to face structured interviews was conducted after 4weeks of intervention to explore the effectiveness of median nerve mobilization on reduction of spasticity and the improvement of upper limb strength.

DETAILED DESCRIPTION:
Spasticity after stroke is common that affect upper limb strength and make activities of daily living difficult. There are many techniques but not any standardized technique for long term effect on reduction of spasticity and improving upper limb strength. This study aimed to explore and understand the effectiveness of neural mobilization on reduction of spasticity and improving upper limb strength in individuals with stroke. This is mixed method approach of embedded design, multicentric study recruited 7 individuals with stroke as no new themes or codes were emerging (data saturated). Median nerve mobilization was given 20 oscillations per minute for 3 times & repeated 3 times with a pause of 1 minute between each sets for 5times/week for 4weeks. Primary outcome measure was Modified Ashworth Scale (MAS) to assess elbow and wrist flexors spasticity and secondary outcome measures were Brunnstrom's stages for hand recovery and Hydraulic hand dynamometer(HHD) to measure grip and pinch strength. Pre and post outcomes data were collected at baseline and 4weeks after intervention and in depth face to face structured interviews was conducted after 4weeks of intervention to explore the effectiveness of median nerve mobilization on reduction of spasticity and the improvement of upper limb strength.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with subacute and chronic stroke (1month and above) having upper limb spasticity.
2. Participants with haemorrhagic and ischemic stroke.
3. Participants who tolerate the supine position.
4. Participants who are oriented and alert.
5. Both males and females.
6. Participants older than 18 years.

Exclusion Criteria:

1. Participants with a score greater than 3 on The Modified Ashworth Scale.
2. Participants with affected speech.
3. Participants with upper limb deformity.
4. Participants experiencing dizziness.
5. Any increase in the dosage of anti-spastic medications during the intervention period.
6. General health problems or pathologies that affect the nervous system like uncontrolled diabetes, hypertension and recent surgeries.
7. Recent onset of worsening neurological signs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-11-22 (Actual); Primary Completion 2022-02-19 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | Change from baseline and 4 weeks
  For spasticity, Total 4 grades are there. Grade 0 means no increase in muscle tone and grade 4 means affected part rigid in flexion or extension. More grade means more spasticity is there.

SECONDARY OUTCOMES:
Brunnstrom's stages for hand recovery | Change from baseline and 4 weeks
  To check recovery of hand functions. Total 7 grades are there. Increase in grade means increase in hand functions.
Hydraulic hand dynamometer | Change from baseline and 4 weeks
  For grip and pinch strength

CONTACTS AND LOCATIONS:
Overall Officials: Rittu Sharma, (MPT), Principal Investigator — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Asir John Samuel, Ph.D, Study Chair — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation; Akanksha Saxena, (Ph.D), Study Director — Maharishi Markandeshwar Institute of Physiotherapy and Rehabilitation
Locations (3):
- India (3):
  - Maharishi Markandeshwar Institute of Physiotherapy & Rehabilitation, Ambāla, Haryana
  - Healing Hands Physiotherapy & Rehabilitation, Hisar, Haryana
  - Bedi Hospital, Kaithal, Haryana